CLINICAL TRIAL: NCT02820623
Title: Increasing Accuracy and Efficiency of Fidelity Measurement in CBT
Brief Title: Project FACTS (Fidelity Accuracy: Comparing Three Strategies)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Rinad Beidas, Ralph Seal Paffenbarger Professor and Chair, Department of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH108551 (NIH)
Record Dates: First submitted 2016-06-03; First posted 2016-07-01 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Assess Fidelity to Cognitive-behavioral Therapy for Youth
Keywords: implementation; fidelity; cognitive behavioral therapy
MeSH Terms: interventions — Self Report

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Self-report (Experimental): Therapists randomized to this condition will complete a brief self-report measure, the Therapy Process Observational Coding System for Child Psychotherapy Strategies Scale-Self Report version (TPOCS-SR) for each of the recorded clinical encounters with enrolled youth. The TPOCS-SR will be a self-report version of the Therapy Process Observational Coding System for Child Psychotherapy-Strategies Scale (TPOCS-S) and will be created in collaboration with the instrument developer (McLeod). In this condition, the investigators will (a) provide an operational definition for each item on the TPOCS-SR (e.g., cognitive education: teaches client the cognitive model (e.g., thoughts influence behavior)/identifies how the cognitive model applies to a specific aspects of the client's life), and (b) provide therapists with a 30-minute training session that includes sample vignettes of particular behaviors and information about how those vignettes should be rated.
  Interventions: Behavioral: Self-report
- Chart Stimulated Recall (Experimental): Therapists randomized to this condition will be asked to bring the charts of three enrolled youth to the chart-stimulated recall interview. A trained interviewer will ask the therapists how well they recall the encounter (rating of memory quality) followed by an open-ended question ("Talk me through your last session with your client. Tell me what you did."). While the therapists are speaking, the interviewer will note any elements that represent a prescribed CBT strategy. The interviewer will go through a list of cognitive-behavioral strategies based upon the TPOCS-S and probe to determine if the therapists completed any of the strategies. Follow-up questions will be used to explore to what degree an element was used and how skillfully and responsively the strategies were used.
  Interventions: Behavioral: Chart-Stimulated Recall
- Behavioral Rehearsal (Experimental): Therapists randomized to this condition will be asked to engage in role-plays demonstrating the CBT strategies used with the three enrolled youth. The investigators will provide therapists with a list of the TPOCS-S CBT strategies and ask them to identify the CBT strategies used in their recorded encounter. The investigators will randomly select one of the strategies they report for each role-play. The investigators will then tell them, "Please role-play how you used this strategy in session with your client, with the trained actor in front of you." Later, an independent rater will rate therapists' adherence and skill based on established scoring criteria.
  Interventions: Behavioral: Behavioral Rehearsal

INTERVENTIONS:
Behavioral: Self-report
  Arms: Self-report
Behavioral: Chart-Stimulated Recall
  Arms: Chart Stimulated Recall
Behavioral: Behavioral Rehearsal
  Arms: Behavioral Rehearsal

SUMMARY:
The objective is to compare the accuracy, costs, and cost-effectiveness of three fidelity measurement methods to assess fidelity to cognitive-behavioral therapy for youth. The investigators will randomize 135 therapists, implementing cognitive-behavioral therapy, to 3 conditions: self-report, chart stimulated recall, and behavioral rehearsal (N = 45 for each group). To calculate the outcomes of interest, each condition will be compared to the gold-standard fidelity measurement method, direct observation.

DETAILED DESCRIPTION:
To achieve the primary objective, the investigators plan to (1) identify the most accurate fidelity measurement method; (2) estimate the economic costs and cost-effectiveness of the fidelity measurement methods; and (3) compare stakeholders' motivation to use each method, as well as identify their perceived barriers and facilitators to use of each method. This study will have a significant positive impact in two ways. First, it will validate fidelity measurement methods that can be used for research. Second, it will produce tools that can be used by community mental health clinics to monitor therapist fidelity, an indicator of therapy quality.

ELIGIBILITY:
Inclusion Criteria: Therapists

* they provide mental health treatment services in community mental health agencies in the City of Philadelphia participating in this study and

  * have been trained in cognitive-behavioral therapy (CBT) through the City-sponsored CBT evidence-based practice initiatives, and/or
  * respond to a brief screening survey that they use CBT; and/or
  * are nominated by a supervisor as a therapist who uses CBT.

Exclusion Criteria: Therapists

* n/a

Inclusion Criteria: Supervisors

* they are supervisors or administrators (i.e., they hold leadership positions) in community mental health agencies in the City of Philadelphia participating in this study.

Exclusion Criteria: Supervisors

* n/a

Inclusion Criteria: Youth and their Legal Guardians

* Youth and their legal guardians will be eligible to participate in this study if the youth

  * is 3-24 years old and
  * has completed at least one session with a therapist who has enrolled to participate in this study.

Exclusion Criteria: Youth and their Legal Guardians

* if the child does not have a legal guardian who is able to consent (e.g., the Department of Human Services (DHS) is the guardian).

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-11; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rinad S Beidas, PhD, Principal Investigator — Northwestern University; Emily M Becker-Haimes, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Becker-Haimes EM, Marcus SC, Klein MR, Schoenwald SK, Fugo PB, McLeod BD, Dorsey S, Williams NJ, Mandell DS, Beidas RS. A Randomized Trial to Identify Accurate Measurement Methods for Adherence to Cognitive-Behavioral Therapy. Behav Ther. 2022 Nov;53(6):1191-1204. doi: 10.1016/j.beth.2022.06.001. Epub 2022 Jun 10. PMID 36229116
- [Derived] Beidas RS, Maclean JC, Fishman J, Dorsey S, Schoenwald SK, Mandell DS, Shea JA, McLeod BD, French MT, Hogue A, Adams DR, Lieberman A, Becker-Haimes EM, Marcus SC. A randomized trial to identify accurate and cost-effective fidelity measurement methods for cognitive-behavioral therapy: project FACTS study protocol. BMC Psychiatry. 2016 Sep 15;16(1):323. doi: 10.1186/s12888-016-1034-z. PMID 27633780

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 126 therapists in the study; these participants consented and were randomized to treatment.
  We assessed 304 therapists for enrollment in the study; of the therapists who were not enrolled, 86 did not meet inclusion criteria, 84 declined to participate, and 8 were excluded for other reasons.
Groups:
- Self-report: Therapists randomized to this condition will complete a brief self-report measure, the Therapy Process Observational Coding System for Child Psychotherapy Strategies Scale-Self Report version (TPOCS-SR) for each of the recorded clinical encounters with enrolled youth. The TPOCS-SR will be a self-report version of the Therapy Process Observational Coding System for Child Psychotherapy-Strategies Scale (TPOCS-S) and will be created in collaboration with the instrument developer (McLeod). In this condition, the investigators will (a) provide an operational definition for each item on the TPOCS-SR (e.g., cognitive education: teaches client the cognitive model (e.g., thoughts influence behavior)/identifies how the cognitive model applies to a specific aspects of the client's life), and (b) provide therapists with a 30-minute training session that includes sample vignettes of particular behaviors and information about how those vignettes should be rated.
  Self-report
- Chart Stimulated Recall: Therapists randomized to this condition will be asked to bring the charts of three enrolled youth to the chart-stimulated recall interview. A trained interviewer will ask the therapists how well they recall the encounter (rating of memory quality) followed by an open-ended question ("Talk me through your last session with your client. Tell me what you did."). While the therapists are speaking, the interviewer will note any elements that represent a prescribed cognitive behavioral therapy (CBT) strategy. The interviewer will go through a list of cognitive-behavioral strategies based upon the TPOCS-S and probe to determine if the therapists completed any of the strategies. Follow-up questions will be used to explore to what degree an element was used and how skillfully and responsively the strategies were used.
  Chart-Stimulated Recall
- Behavioral Rehearsal: Therapists randomized to this condition will be asked to engage in role-plays demonstrating the CBT strategies used with the three enrolled youth. The investigators will provide therapists with a list of the TPOCS-S CBT strategies and ask them to identify the CBT strategies used in their recorded encounter. The investigators will randomly select one of the strategies they report for each role-play. The investigators will then tell them, "Please role-play how you used this strategy in session with your client, with the trained actor in front of you." Later, an independent rater will rate therapists' adherence and skill based on established scoring criteria.
  Behavioral Rehearsal
Period: Overall Study
Arm/Group | Self-report | Chart Stimulated Recall | Behavioral Rehearsal
Started | 41 | 42 | 43
Completed | 36 | 35 | 32
Not Completed | 5 | 7 | 11
Not completed — Withdrawal by Subject | 1 | 3 | 3
Not completed — Participation interrupted due to COVID-19 | 3 | 3 | 2
Not completed — Therapist unable to enroll clients | 1 | 1 | 3
Not completed — Clients declined, piloting condition, or only telehealth | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Chart Stimulated Recall: Therapists randomized to this condition will be asked to bring the charts of three enrolled youth to the chart-stimulated recall interview. A trained interviewer will ask the therapists how well they recall the encounter (rating of memory quality) followed by an open-ended question ("Talk me through your last session with your client. Tell me what you did."). While the therapists are speaking, the interviewer will note any elements that represent a prescribed CBT strategy. The interviewer will go through a list of cognitive-behavioral strategies based upon the TPOCS-S and probe to determine if the therapists completed any of the strategies. Follow-up questions will be used to explore to what degree an element was used and how skillfully and responsively the strategies were used.
  Chart-Stimulated Recall
- Total: Total of all reporting groups
Arm/Group | Self-report | Chart Stimulated Recall | Behavioral Rehearsal | Total
Number analyzed (Participants) | 41 | 42 | 43 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number of participants analyzed for each group does not match overall number of baseline participants in that group because some participants did not disclose their age.
  years
    number analyzed (Participants) | 40 | 40 | 42 | 122
    (all) | 39.93 (13.81) | 37.42 (12.13) | 34.76 (11.76) | 37.33 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number of participants analyzed for each group does not match overall number of baseline participants in that group because some participants did not disclose their sex.
  Participants
    number analyzed (Participants) | 40 | 40 | 42 | 122
    Female | 25 | 32 | 37 | 94
    Male | 15 | 8 | 5 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6 | 12
  Not Hispanic or Latino | 36 | 37 | 37 | 110
  Unknown or Not Reported | 2 | 2 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 5 | 6 | 22
  White | 23 | 32 | 29 | 84
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 6 | 3 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 41 | 42 | 43 | 103
Education [Count of Participants; unit: Participants] — Population: Number of participants analyzed for each group (for some group[s[) does not match overall number of baseline participants in that group (for some group[s]) because some participants did not disclose their level of education.
  Participants
    number analyzed (Participants) | 41 | 40 | 43 | 124
    Bachelor's Degree | 0 | 2 | 2 | 4
    Master's Degree | 40 | 37 | 39 | 116
    Doctorate | 1 | 1 | 2 | 4
Years Experience [Mean (Standard Deviation); unit: years] — Population: Number of participants analyzed for one or more group(s) does not match overall number of baseline participants in that group(s) because some participants did not disclose their number of years' experience.
  years
    number analyzed (Participants) | 41 | 40 | 43 | 124
    (all) | 11.44 (10.57) | 10.55 (10.29) | 8.12 (9.76) | 10.00 (10.22)
Type of Employee [Count of Participants; unit: Participants]
  Salaried | 22 | 20 | 22 | 64
  Fee for service | 18 | 18 | 18 | 54
  No response | 1 | 4 | 3 | 8
Participated in city sponsored Evidence-Based Practice training initiative [Count of Participants; unit: Participants] | 29 | 25 | 28 | 82
Number of client sessions recorded in the study [Mean (Standard Deviation); unit: sessions] | 2.44 (1.05) | 2.29 (1.17) | 2.14 (1.32) | 2.29 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: Total Fidelity Scores for Each Study Condition Measured Via Direct Observation (TPOCS-RS) and Study Arm Fidelity Method Scores
Description: Client sessions for all 3 conditions were scored for CBT adherence via direct observation using the Therapy Process Observational Coding System-Revised Strategies (TPOCS-RS) Scale (McLeod et al., 2015) on a 7-point Likert Scale (1='not at all,' 7='extensively'). We analyzed the TPOCS-RS' Maximum CBT score (highest coded intervention technique across all 12 possible interventions in a given session).
  We also measured CBT adherence during client sessions using the strategies from each study condition (described in 'Arms/Groups' below). All 3 conditions used parallel 7-point scales to the TPOCS-RS.
  Higher scores for the 3 study condition strategies indicate greater reported use, and higher scores on the TPOCS-RS indicate greater observed use of CBT interventions. Our goal was to compare the study condition methods of assessing CBT adherence to direct observation (TPOCS-RS), the gold standard.
Time Frame: through study completion, an average of 1 month
Population: Participants (i.e., therapists) were assigned to one of 3 conditions: self-report, chart stimulated recall, or behavioral rehearsal. The unit of analysis for Maximum Mean condition score and Maximum Mean direct observation (TPOCS-RS) score was client session; therapists could include more than one client session for inclusion in analyses.
Measure: Mean (Standard Deviation); unit: Maximum CBT score on a scale
Units Other Than Participants: Client Sessions
Arm/Group | Self-report | Chart Stimulated Recall | Behavioral Rehearsal
Number analyzed (Participants) | 41 | 42 | 43
Number analyzed (Client Sessions) | 100 | 96 | 92
Maximum CBT score on a scale
  Maximum Mean Condition Score | 5.28 (1.17) | 4.53 (1.18) | 4.09 (1.48)
  Maximum Mean direct observation (TPOCS-RS) Score | 3.42 (1.55) | 3.69 (1.36) | 3.72 (1.59)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from study initiation through study completion, an average of 6 weeks for each participant.
Arm/Group | Self-report | Chart Stimulated Recall | Behavioral Rehearsal
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/41 | 0/42 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT02820623/Prot_SAP_000.pdf